CLINICAL TRIAL: NCT05650060
Title: The Characteristics of Patients Treated With Secukinumab for Moderate to Severe Plaque Psoriasis in Real-world Practice in Thailand
Brief Title: Characteristics of Patients Treated With Secukinumab for Moderate to Severe Plaque Psoriasis
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457ATH01
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Plaque Psoriasis
Keywords: secukinumab,; psoriasis,; effectiveness,; real-world,; Thailand
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Secukinumab: all patients with psoriasis who received secukinumab
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — all patients with psoriasis who received secukinumab

SUMMARY:
This study was a non-interventional, retrospective study collecting data from hospital medical records. Approximately 200 adult patients with moderate to severe plaque psoriasis who were treated with secukinumab from hospitals in Thailand that participated in this study were expected for data collection.

DETAILED DESCRIPTION:
The study was performed in 7 study sites in Thailand and planned to involve approximately 200 medical records.

At each study site, patients who were treated with secukinumab or had ever been treated with secukinumab for moderate to severe plaque psoriasis were included for screening by chronological order starting from the most recent date (April 2021) to September 2017. This was to include the most recent clinical practice in the study.

The data of patients diagnosed with moderate-to-severe chronic plaque-type psoriasis who received secukinumab in real clinical practice at least 1 dose were collected. The medical records were reviewed to collect the data from the date of the first diagnosis of psoriasis till the most recent dose of secukinumab.

The data of secukinumab use and clinical outcome (PASI score) were collected at 4 and 16 weeks after first dose initiation and at the most recent dose of secukinumab. The total number of secukinumab injections at the 3-time points were collected.

An index date was defined for each patient. The first secukinumab injection observed in the medical records was considered the index date for the exploratory endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female aged ≥ 18 years at index date
* Previous diagnosis of moderate to severe plaque psoriasis as hospital record with available baseline PASI at index date (date 0 to date -7 prior index date)
* Initiated treatment with secukinumab for moderate to severe plaque psoriasis during September 2017-April 2021

Exclusion Criteria:

- Patients diagnosed with other forms of psoriasis other than plaque-type

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was a retrospective medical chart review study. It collected the characteristics of patients who received secukinumab for the treatment of moderate to severe plaque psoriasis as the primary objective.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Age | Baseline
  Age information was reported.
Gender | Baseline
  Gender information was reported.
Number of patients with Reimbursement scheme | Baseline
  Reimbursement scheme information was reported.
Weight | During 3 months pre-baseline
  Weight information was reported.
Height | During 3 months pre-baseline
  Height information was reported.
BMI | During 3 months pre-baseline
  BMI information was reported.
Co-morbidities | During 12 months pre-baseline
  * Crohn's Disease
  * Diabetes Mellitus
  * Dyslipidemia
  * Hypertension
  * Inflammatory Bowel Disease
  * Latent Tuberculosis
  * Psoriatic Arthritis (PsA)
Psoriasis Area and Sensitivity Index (PASI) score | During 4 weeks pre-baseline
  Psoriasis Area and Severity Index (PASI) is the most widely used tool for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease).
Percentage of Body Surface Area (BSA) involvement | During 4 weeks pre-baseline
  Percentage of Body Surface Area (BSA) involvement was reported.
Disease Life Quality Index (DLQI) score | During 4 weeks pre-baseline
  The Dermatology Life Quality Index (DLQI) is a simple, self-administered and user-friendly validated questionnaire. The DLQI is designed to measure the health-related quality of life of adult patients suffering from a skin disease. The DLQI is a validated, 10-question, self-reported questionnaire to evaluate the patient's perception of the impact of psoriasis on quality of life. The DLQI was rated on a 4-point scale (0 = not at all to 3 = very much). The highest possible total score for the DLQI is 30 and higher scores indicate more severe impact on quality of life.
Date of first symptom of psoriasis (PSO) / year | Approximately 2 years pre-baseline (PSO diagnosed date to index date, where index date is defined as date of initiation of treatment)
  To describe the PSO treatment history
Date of psoriasis diagnosis / year | Approximately 2 years pre-baseline (PSO diagnosed date to index date, where index date is defined as date of initiation of treatment)
  To describe the PSO treatment history
Duration of psoriasis diagnosis | Approximately 2 years pre-baseline (PSO diagnosed date to index date, where index date is defined as date of initiation of treatment)
  To describe the PSO treatment history
Date of first systemic treatment/ year | Approximately 2 years pre-baseline (PSO diagnosed date to index date, where index date is defined as date of initiation of treatment)
  To describe the PSO treatment history
Date of first biologic agent/year | Approximately 2 years pre-baseline (PSO diagnosed date to index date, where index date is defined as date of initiation of treatment)
  To describe the PSO treatment history
Duration of topical therapy | Approximately 2 years pre-baseline (PSO diagnosed date to index date, where index date is defined as date of initiation of treatment)
  To describe the PSO treatment history
History of topical therapy | Approximately 2 years pre-baseline (PSO diagnosed date to index date, where index date is defined as date of initiation of treatment)
  To describe the PSO treatment history
Duration of systemic therapy | Approximately 2 years pre-baseline (PSO diagnosed date to index date, where index date is defined as date of initiation of treatment)
  To describe the PSO treatment history
History of systemic therapy | Approximately 2 years pre-baseline (PSO diagnosed date to index date, where index date is defined as date of initiation of treatment)
  To describe the PSO treatment history
Duration of biologic therapy | Approximately 2 years pre-baseline (PSO diagnosed date to index date, where index date is defined as date of initiation of treatment)
  To describe the PSO treatment history
History of biologic therapy | Approximately 2 years pre-baseline (PSO diagnosed date to index date, where index date is defined as date of initiation of treatment)
  To describe the PSO treatment history
Date of PsA diagnosis/year | Approximately 2 years pre-baseline (PSO diagnosed date to index date, where index date is defined as date of initiation of treatment)
  To describe the PSO treatment history
Duration of PsA diagnosis | Approximately 2 years pre-baseline (PSO diagnosed date to index date, where index date is defined as date of initiation of treatment)
  To describe the PSO treatment history
Number of patients with baseline PSO treatment | During 12 months pre-baseline
  Topical Therapies
  * Topical corticosteroid
  * Coal tar
  * Salicylic acid
  * Vitamin D analogues
  * Anthralin
  * Calcineurin inhibitors
  * Others Oral systemic therapies
  * Methotrexate
  * Acitretin
  * Retinoid
  * Cyclosporine
  * Azathioprine
  * Hydroxyurea
  * Leflunomide
  * Sulfasalazine
  * Others Biologic therapy
  * Infliximab
  * Etanercept
  * Ustekinumab
  * Brodalumab
  * Guselkumab
  * Ixekizumab
  * Others
Duration since the discontinuation of the latest biological agents | Baseline
  Secukinumab therapy
Medication use concomitant to index secukinumab prescription | Baseline
  Secukinumab therapy
Treatment pattern with secukinumab | Baseline
  Secukinumab therapy
Treatment duration since the first dosing till the most recent dosing | Baseline
  Secukinumab therapy

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No